CLINICAL TRIAL: NCT06385574
Title: The Effects of Technological Based Rehabilitation on Individuals With Rheumatic Disease With Hand Involvement
Brief Title: Technological Based Rehabilitation on Individuals With Rheumatic Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sebahat Yaprak Cetin, PT, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-088
Record Dates: First submitted 2024-04-22; First posted 2024-04-26 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Rheumatic Diseases; Hand Rheumatism; Virtual Reality Therapy
Keywords: rheumatic diseases; hand exercises; leap motion; functionality
MeSH Terms: conditions — Rheumatic Diseases | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Intervention Model Description: There are three groups in the study. First group is leap motion interventional group, second group is hand exercises group and the third group is waiting list.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcome assessors do not know which patient is in which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality therapy group (Experimental): Individuals in this group will be given hand exercises (wrist flexion, extension and deviations) for 45 minutes, 2 days a week for 8 weeks, using a leap motion control device and games selected in accordance with this device.
  Interventions: Other: Virtual reality therapy
- Conventional exercise group (Experimental): Hand exercises (wrist flexion, extension and deviations)) will be applied to individuals in this group under the supervision of a specialist physiotherapist for 45 minutes, 2 days a week for 8 weeks.
  Interventions: Other: Virtual reality therapy
- Control group (No Intervention): This group is waiting list. After the study, patients will do hand exercises with the leap motion controller device.

INTERVENTIONS:
Other: Virtual reality therapy — Conventional hand therapy
  Other Names: Hand exercises
  Arms: Conventional exercise group; Virtual reality therapy group

SUMMARY:
Affects such as pain, swelling, tenderness, deformities, limitations, strength and function losses, skill and coordination deficiencies in the hand joints, which are frequently seen in rheumatism patients with hand involvement, are included in body structure and function disorders within the framework of International Classification of Function System. Leap Motion Controller is used in hand rehabilitation because it is small in size, low-cost, portable, non-contact, easy to use and provides visual and auditory feedback. The aim of our study is to examine the effect of technology-based rehabilitation on joint range of motion, grip strength, functionality and disease activity in adult individuals with rheumatic disease with hand involvement; and also to compare these effects with the effects of the hand rehabilitation program implemented under the guidance of a physiotherapist and the control group that continues its routine life.

DETAILED DESCRIPTION:
In the study, 45 adult individuals diagnosed with rheumatic disease with hand involvement will be randomly divided into 3 groups. The first group will be given virtual reality exercises via Leap Motion Controller. Virtual reality exercises will be applied 30 minutes a day, 3 days a week for 8 weeks. To the second group, a conventional hand rehabilitation program will be applied under the supervision of a physiotherapist. The hand rehabilitation program will be applied 30 minutes a day, 3 days a week for 8 weeks. The third group will be the control group, which continues with its routine medications and is not included in any exercise program. After randomization, the individuals' joint range of motion, gross and fine grip strength, functionality, and disease activities will be evaluated. Evaluations will be made twice, at the beginning and at the end of the 8-week program. Disease Activity Score 28 (DAS 28), hand dynamometer, picnometer, Jebsen Hand Function Test, Nine Hole Peg Test, Duruoz Hand Index and Michigan Hand Outcome questionnairre will be used for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with a rheumatic disease that meets the latest criteria by a rheumatologist
* Involvement in hand joints (pain, swelling, tenderness)
* Being 18 years or older
* Being on stable drug treatment for the last 6 months
* Having sufficient cooperation to participate in the study
* Volunteering to participate in the study

Exclusion Criteria:

* Not volunteering to participate in the study
* Having difficulty in cooperating at work
* Having an additional orthopedic and/or neurological disease that will affect hand functions

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Hand grip strength measurement | 8 weeks
  Hand grip strength will be measured with a Jamar hydraulic hand dynamometer. Grip tests will be performed in the standard position recommended by the American Association of Hand Therapists. This is the standard position; The patient will be seated in a position that provides 90-20 degree flexion of the hip and knee, shoulder adduction, forearm neutral position, 90 degree flexion of the elbow, 0-30 degree extension of the wrist and 0-15 degree ulnar deviation. The measurement will be repeated three times. There will be a 15-second rest break at the end of each measurement. As a result, the average of three measurements will be recorded.
Jebsen Hand Function Test (JHFT) | 8 weeks
  This test consists of tasks involving grasping types commonly used in daily living activities and evaluates people's speed in these tasks. Each stage of the Jebsen Taylor Hand Function Test, which consists of seven sub-steps, will be explained to the individuals in detail before the task and the individuals will be asked to try the task. Estimated time to complete 7 subtasks is 20 minutes. Individuals will complete tasks with both their dominant and non-dominant hands. The task will start with the practitioner's "start" command, and when the task is completed, the test performance will be recorded separately for the tested hand as the time to complete the task. Below is the tasks.
  Task 1: Stack 4 checkers, Task 2: Card flipping, Task 3: Collecting objects, Task 4: Writing,Task 5: Eating, Task 6: Moving Light Objects, Task 7: Moving Heavy Objects
Nine Hole Peg Test (NHPT) | 8 weeks
  This device is a device consisting of a square platform and a storage box. There are 9 holes in the square-shaped area (12.7x2cm) and 9 cylinders suitable for these holes. The diameter of the holes is 0.71 cm, the diameter of the cylinders is 0.64 cm, the length is 3.2 cm, the distance between the holes is 3.2 cm, the hole depth is 1.3 cm and the size of the storage box is 13x13 cm. During the test, the patient sits at the table with the 9-hole board, and the patient is asked to quickly take the 9 cylinders from the storage box, place them in the holes in random order, and quickly remove them from the holes without taking a break and place them in the storage box. Meanwhile, time is measured in seconds with a stopwatch. The test is performed 2 times consecutively for both hands and the average of the result is taken. The total test score is calculated by taking the average of the scores for both hands.
Duruoz Hand Index (DHI) | 8 weeks
  The test consists of 18 questions. It is a simple, useful and reliable test that is presented by separating daily life functions (kitchen, clothing, cleaning, workplace and other daily life activities), does not require additional training and equipment for the test, and takes approximately 2-3 minutes to apply. It is a simple and understandable test in which questions are answered according to a Likert scale, with a minimum score of 0 and a maximum of 90 points. A lower score indicates a better functional state.
Michigan Hand Outcome questionnaire (MHQ) | 8 weeks
  This questionnaire is a scale consisting of six sections and 57 different items. It helps us question how well patients perform tasks they frequently perform. The patient answers the questions according to the Likert measurement method, which gives values from one to five. Each of the 6 different categories in the scale is scored uniquely. High scores indicate good functionality.

SECONDARY OUTCOMES:
Disease Activity Score 28 (DAS 28) | 8 weeks
  It includes swelling and tenderness in 28 joints including the proximal interphalangeal joint, metacarpophalangeal joint, wrist, elbow, shoulder and knee joints, erythrocyte sedimentation rate (ESR) value, and global evaluation of the patient (VAS 0-100 mm). The DAS 28 value is calculated using a special formula:
  DAS28 = (0.56 x √ Number of Tender Joints) + (0.28 x √ Number of Swollen Joints) + (0.70 x Ln (ESR value)) + (0.014 x Patient global assessment) High score; indicates high disease activity. Values higher than 5.1 indicate high disease activity, values between 3.2<DAS28≤5.1 indicate medium disease activity, values of 2.6<DAS28≤3.2 indicate low disease activity, and values less than or equal to 2.6 indicate that the patient is in remission.
Hand fine grip strength measurement | 8 weeks
  Fine grip strength measurements will be made with finger dynamometry. Grip tests will be performed in the standard position recommended by the American Association of Hand Therapists. This is the standard position; The patient will be seated in a position that provides 90 degrees of hip and knee flexion, shoulder adduction, forearm neutral position, 90 degree flexion of the elbow, 0-30 degree extension of the wrist and 0-15 degree ulnar deviation. Three different finger grips will be evaluated. These:
  1- Fingertip grip strength, 2- Lateral grip strength, 3- Three point grip strength.
  Measurements will be repeated three times. There will be a 15-second rest break at the end of each measurement. As a result, the average of three measurements will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sebahat Yaprak Cetin, PhD, Principal Investigator — Akdeniz University
Locations (1):
- Sebahat Yaprak Cetin, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will share data to the other individuals with some analyses program.